CLINICAL TRIAL: NCT06931288
Title: Study on the Effectiveness of Atrial Fibrillation Screening Using Electronic Blood Pressure Monitor With Atrial Fibrillation Detection Function
Brief Title: Electronic Blood Pressure Monitor for Atrial Fibrillation Detection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AFSE
Record Dates: First submitted 2025-04-01; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Detection; Electronic blood pressure monitor
MeSH Terms: conditions — Atrial Fibrillation | interventions — Blood Pressure Monitors

STUDY DESIGN:
Intervention Model Description: The eligible center as a cluster will be randomly assigned to either the single-lead ECG group or the electronic blood pressure monitor group for atrial fibrillation detection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-lead ECG (Active Comparator)
  Interventions: Device: Single-lead ECG
- Blood pressure monitor (Experimental)
  Interventions: Device: Blood pressure monitor

INTERVENTIONS:
Device: Blood pressure monitor — In the trial group, atrial fibrillation screening will be integrated into blood pressure measurements using the BP77A1T electronic blood pressure monitor (Omron Healthcare, Kyoto, Japan).
  Arms: Blood pressure monitor
Device: Single-lead ECG — In the control group, a single-lead ECG will be recorded for 30s with a handheld ECG for atrial fibrillation detection. Each ECG rhythm strip will be reviewed and analyzed by a cardiologist from the research team.
  Arms: Single-lead ECG

SUMMARY:
Study name: Study on the Effectiveness of Atrial Fibrillation Screening Using Electronic Blood Pressure Monitor with Atrial Fibrillation Detection Function

Objective: This study compares an electronic blood pressure monitor (BP77A1T, Omron Healthcare, Kyoto, Japan) with single-lead electrocardiography for atrial fibrillation detection in an elderly Chinese population.

Study design: This study is a cluster-randomized and controlled trial.

Study population: Men and women aged over 60 years meeting the inclusion/exclusion criteria.

Randomization and treatment: Eligible centers as clusters will be randomly assigned to either the single-lead electrocardiography group or the electronic blood pressure monitor group for atrial fibrillation detection.

Sample size: About 50 centers, at least 20,000 participants.

Timeline: Participants enrollment are expected to be performed from May 2025 to July 2026.

Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

DETAILED DESCRIPTION:
Study name: Study on the Effectiveness of Atrial Fibrillation Screening Using Electronic Blood Pressure Monitor with Atrial Fibrillation Detection Function

Rationale: With the advancement of technology and the development of artificial intelligence, it has become possible to detect atrial fibrillation during routine blood pressure measurements. Previous studies have explored the accuracy of the blood pressure monitor for atrial fibrillation detection. However, the efficiency and adherence of using this device for large-scale population screening remain unknown.

Objective: This study compares an electronic blood pressure monitor (BP77A1T, Omron Healthcare, Kyoto, Japan) with single-lead electrocardiography for atrial fibrillation detection in an elderly Chinese population.

Study design: This study is a cluster-randomized and controlled trial. The eligible center as a cluster will be randomly assigned to either the single-lead electrocardiography group or the electronic blood pressure monitor group for atrial fibrillation detection.

Study population: Men and women aged over 60 years meeting the inclusion/exclusion criteria. Inclusion criteria included: 1) Signed and dated informed consent form. 2) Age ≥ 60 years. 3) Able to cooperate with atrial fibrillation screening, complete questionnaires, and communicate normally. The only exclusion criteria is severe communication problem.

Randomization and treatment: Eligible centers as clusters will be randomly assigned to either the single-lead electrocardiography group or the electronic blood pressure monitor group for atrial fibrillation detection. In the control group, a single-lead electrocardiography will be recorded for 30s with a handheld electrocardiography for atrial fibrillation detection. Each ECG rhythm strip will be reviewed and analyzed by a cardiologist from the research team. In the trial group, atrial fibrillation screening will be integrated into blood pressure measurements using the BP77A1T electronic blood pressure monitor (Omron Healthcare, Kyoto, Japan).

Sample size: About 50 centers, at least 20,000 participants.

Timeline: Participants enrollment are expected to be performed from May 2025 to July 2026.

Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form.
2. Age ≥ 60 years.
3. Able to cooperate with atrial fibrillation screening, complete questionnaires, and communicate normally.

Exclusion Criteria:

1. Participants with severe communication problems.

Ages: 60 Years to 125 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2025-05-06 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The difference in detection rates of atrial fibrillation between the blood pressure monitor and the single-lead ECG group. | Baseline

SECONDARY OUTCOMES:
The difference in detection rates atrial fibrillation of between the blood pressure monitor and the single-lead ECG group among screening-positive participants. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai 200025, Shanghai, Shanghai Municipality, China